CLINICAL TRIAL: NCT04783701
Title: Coronary CT Angio Evaluating Graft Patency in ACS Patients Treated With DAPT or Single ASA After CABG (CoCAP)
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Jonas Holm, MD, PhD, University Hospital, Linkoeping
Other Study IDs: CoCAP
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Acute Coronary Syndrome; Coronary Bypass Stenosis
Keywords: Acute coronary syndrome; Coronary bypass surgery; Coronary computed tomography angiography; Antiplatelet therapy
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to compare the presence of graft patency in single aspirin vs dual anti platelet therapy (DAPT) treatment including ticagrelor in patients with acute coronary syndrome (ACS) treated with coronary artery bypass surgery (CABG). Follow up time is 12-36 months postoperatively and the patency will be evaluated with coronary computed tomography angiography (CCTA)

ELIGIBILITY:
Inclusion Criteria:

* Previously included in TACSI-trial

Exclusion Criteria:

* Highly irregular heart rhythm (i.e. atrial fibrillation)
* Chronic kidney disease with estimated glomerular filtration rate (eGFR) <45ml/min/1,73m2
* Body weight >120 kg
* Previous severe allergic reaction (i.e. anaphylactic reaction) to iodine-based contrast agents
* Not able to communicate
* Not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients previously included in the TACSI-trial (Dual antiplatelet therapy with ticagrelor and ASA vs. ASA alone after coronary artery bypass grafting in patients with acute coronary syndrome) . This means patients with age ≥18 years that has undergone for the first time an isolated CABG due to an episode of an acute coronary syndrome (ACS) event within 6 weeks before CABG. The randomized, controlled trial TACSI (ClinicalTrials.gov NCT03560310) offers a unique possibility to address the issue of graft patency based on antiplatelet strategy in patients with acute coronary syndromes.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Graft patency after CABG | 12-36 months
  Defined as patency on CCTA (FitzGibbon A) without previous graft failure identified on CCTA and/or invasive coronary angio (ICA) since CABG, intention to treat (ITT) analysis.

SECONDARY OUTCOMES:
Graft patency after CABG - PP analysis | 12-36 months
  Defined as patency on CCTA (FitzGibbon A) without previous graft failure identified on CCTA and/or ICA since CABG, per protocol (PP) analysis.
Graft patency after CABG | 12-36 months
  Defined as non-occlusion on CCTA (FitzGibbon A+B) without previous graft occlusion identified on CCTA and/or ICA since CABG, ITT analysis.
Graft patency after CABG | 12-36 months
  Defined as non-occlusion on CCTA (FitzGibbon A+B) without previous graft occlusion identified on CCTA and/or ICA since CABG, PP analysis.
Graft patency after CABG | 12-36 months
  Defined as patency on CCTA (FitzGibbon A) without graft failure identified on CCTA and/or ICA since CABG, patients on oral anticoagulants excluded, ITT (sensitivity analysis).
Graft patency after CABG | 12-36 months
  Defined as non-occlusion on CCTA (FitzGibbon A) without previous graft failure identified on CCTA and/or ICA since CABG, patients on oral anticoagulants excluded, PP (sensitivity analysis).

OTHER OUTCOMES:
Subgroup analyses | 12-36 months
  Possible interactions in response to study treatment, with special focus on the following factors; age, gender, renal function, diabetes, oral anticoagulant therapy, adherence to study treatment and time from end of study medication.
Explorative analyses | 12-36 months
  Performed on the graft patency of internal mammary artery (IMA) in the two treatment groups, as well as if there are any differences in graft patency between different anastomoses and grafting techniques.
  Possible predictors of graft failure in general, with age, gender, diabetes, obesity, renal failure, urgency level and length of surgery, per-operative complications, number and type of graft as well as pre-operative fractional flow reserve as variables to explore.
  Gender analysis will be performed, analyzing if female gender is associated with worse prognosis post CABG, adjusting for their higher age and burden of co-morbidities.

CONTACTS AND LOCATIONS:
Locations (6):
- Norway (2):
  - Department of Heart Disease, Haukeland University Hospital, Bergen
  - St Olavs University Hospital, Trondheim
- Sweden (4):
  - Department of Molecular and Clinical Medicine, Wallenberg Laboratory, Institute of Medicine, Gothenburg
  - Dep of Vascular and Thoracic Surgery, Örebro
  - Department of Cardiothoracic Surgery Karolinska University Hospital, Stockholm
  - University Hospital Linköping, Linköping, Östergötland County